CLINICAL TRIAL: NCT05110313
Title: Effects of Tildrakizumab (ILUMYA) Use on Epigenetic Age Acceleration and Psoriasis
Brief Title: Effects of Tildrakizumab on Epigenetic Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carlos Wambier (Other)
Collaborators: Sun Pharmaceutical Industries Limited (Industry); Brown University (Other); Lifespan (Other); Ocean State Research Institute, Inc. (Other)
Responsible Party: Sponsor-Investigator, Carlos Wambier, Associate Professor of Dermatology, Clinician Educator, Rhode Island Hospital
Organization: Rhode Island Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 420620; 20-056 (Other: Study ID Rhode Island Hospital)
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Psoriasis; Aging; Epigenetic Disorder; Inflammation; Skin
Keywords: Epigenetic aging; DNA methylation; interleukin (IL)-23; Neutrophilic inflammation; Psoriasis; Aging; Transcriptome
MeSH Terms: conditions — Psoriasis; Dermatitis | interventions — tildrakizumab; World Health Organization

STUDY DESIGN:
Intervention Model Description: We will enroll 30 subjects aged 35 years or older.
  Arm 1 (psoriasis treatment): 20 subjects with moderate-to-severe psoriasis (including 10 men and 10 women).
  Arm 2 (non-psoriasis, non-treatment): 10 age and sex matched controls without psoriasis (including 5 men and 5 women).
  The blood leukocytes will be collected to evaluate DNA methylation at baseline (week 0) for both arms. The psoriasis treatment arm will undergo blood leukocytes collection during treatment (at week 28) and post-treatment (week 52).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PSORIASIS TREATMENT (Experimental): 1 syringe containing 1 mL of 100 mg/mL tildrakizumab-asmn. 100mg delivered by subcutaneous injection at weeks 0, 4, 16 and 28. Total of 20 subjects (10 male, 10 female).
  Interventions: Biological: TILDRAKIZUMAB
- NON-PSORIASIS (No Intervention): No intervention. Total of 10 subjects (5 male, 5 female).

INTERVENTIONS:
Biological: TILDRAKIZUMAB — ILUMYA (tildrakizumab-asmn) is a humanized IgG1/k monoclonal antibody that selectively binds to the p19 subunit of IL-23 and inhibits its interaction with the IL-23 receptor. IL-23 is a naturally occurring cytokine that is involved in inflammatory and immune responses.
  ILUMYA injection for subcutaneous use is a sterile, clear to slightly opalescent, colorless to slightly yellow solution supplied in 1mL single-dose prefilled syringe which contains 100 mg of tildrakizumab-asmn formulated in: L-histidine (0.495 mg), L-histidine hydrochloride monohydrate (1.42 mg), polysorbate 80 (0.5 mg), sucrose (70.0 mg), and Water for Injection, USP with a pH of 5.7-6.3. ILUMYA is supplied in a single-dose prefilled syringe with a glass barrel and 29-gauge fixed, 1/2-inch needle.
  Other Names: ILUMYA™; tildrakizumab-asmn; ATC CODE: L04AC17 (WHO)
  Arms: PSORIASIS TREATMENT

SUMMARY:
Design: Single-center open-label clinical trial.

Objective: Evaluate if tildrakizumab reverses peripheral blood leukocyte DNA methylation (epigenetic aging) observed in chronic psoriasis.

Number of subjects: 30. Intervention group: 20 (10 men, 10 women) with moderate-to-severe psoriasis. Control group: 10 (5 men, 5 women) with other skin diagnosis.

Population: >35-year-old subjects will be recruited from Brown Dermatology clinics.

Biological samples: Blood samples will be collected for all subjects at screening, and weeks 16, 28 and 52. Urine pregnancy tests will be performed for females of childbearing potential at weeks 4, 16, and 28. Serum pregnancy test and QuantiFERON test for tuberculosis will be performed at screening visit.

Safety parameters: Adverse events, and screening, week 16, week 28 blood samples laboratory results. Females of childbearing potential: serum pregnancy test at screening visit, urine pregnancy test at weeks 4, 16, and 28. Data Safety Monitoring Board will review data and laboratory flags quarterly.

Study center: Rhode Island Hospital, Providence, RI, USA.

Trial Duration: One year.

DETAILED DESCRIPTION:
1. Introduction

   Psoriasis is a common, chronic, inflammatory disorder that affects millions of individuals worldwide.1,2 Although psoriasis etiology is still largely unknown and its precision management remains to be improved, advances in understanding the pathogenic cytokine network of psoriasis have led to the development of biologic therapy, such as FDA-approved on-label indication for moderate-to-severe psoriasis of tildrakizumab-asmn (ILUMYA, Sun Pharma Global, Princeton, NJ), an injectable monoclonal antibody that inhibit interleukin (IL)-23, a pro-inflammatory cytokine. Epidemiologic studies have promoted the recognition of psoriasis as a systemic disorder.3 Associations between psoriasis and incident risk of diabetes, cardiovascular disease, Crohn's disease, and gout have been reported in prospective studies.4-7 However, the mechanism underlying the systemic manifestations has been a knowledge gap for research on psoriasis.8
2. Epigenetic aging (DNA methylation)

   The complex interplay of genetic and environmental factors in psoriasis may occur through the epigenetic mechanisms. DNA methylation of cytosine followed by guanine residues (CpG dinucleotides), the epigenetic process that participates in the transcriptional regulation and gene expression, has been linked to psoriasis.9 As the precise pathogenesis underlying the development of psoriasis remains largely undefined, further exploration of the role of epigenetics would offer a biologically plausible perspective to clarify psoriasis etiology. Epigenetic epidemiology would serve as a tool to elucidate the susceptibility and to identify novel biomarkers for psoriasis.10 The epigenetic clock is a novel biomarker of aging, developed based on DNA methylation.11-13 The epigenetic clock may capture aspects of "biological age" and older epigenetic age of blood has been associated with all-cause mortality,14,15 obesity,16 and many diseases.17-20 Although whether epigenetic age is associated with psoriasis is not yet known, previous research from our group recently found that average epigenetic age in psoriasis patients was 5 years higher than their corresponding chronological age (data not published), suggesting possible epigenetic age acceleration in psoriasis. Therefore, epigenetic age acceleration may serve as a novel biomarker for psoriasis and its systemic manifestations. It may also potentially be used as an intermediate biomarker assessing the systemic effects of tildrakizumab.

   Blood-based measures of epigenetics have the advantage of interrogating the systemic health status or treatment responses and assessing biomarkers across a large variety of disease domains.10,21

   Rationale for the study:

   Although epigenetic changes are tissue-specific, the connections between epigenetic epidemiology and psoriasis in blood-based epigenetic studies would decipher novel systemic inflammation and immune states of psoriasis and elucidate the effect of tildrakizumab use on the epigenetic age acceleration. Comprehensive assessment of epigenetic age acceleration in blood leukocytes between psoriasis and controls, and the change in epigenetic age acceleration after tildrakizumab initiation may lead to the identification of methylation markers for predicting the systemic risk of psoriasis and the effect of tildrakizumab on psoriasis. If confirmed to be an intermediate marker for the effect of psoriasis therapy with tildrakizumab, epigenetic age may be used to better profile the beneficial role of immunomodulation, promoting the management of psoriasis and its systemic comorbidities.

   Psoriasis is an inflammatory disease of the skin and joints and has been recognized as a systemic disorder. In this proposed study, the investigators hypothesize that epigenetic age acceleration may be associated with psoriasis, and tildrakizumab may be able to affect the epigenetic age acceleration associated with psoriasis.
3. Objective

To determine the association between epigenetic age acceleration and risk of psoriasis, and also to evaluate if tildrakizumab can reverse peripheral blood leukocyte DNA methylation (epigenetic aging) associated with chronic psoriasis.

Specific Aim 1: To examine the association between epigenetic age acceleration and psoriasis: by comparing the baseline samples of peripheral blood leukocyte genome-wide DNA methylation assay collected at screening for psoriasis patients and controls.

Specific Aim 2: To evaluate dynamic changes in epigenetic age of the on-label use of tildrakizumab (week 28 vs screening visit). And upon discontinuation (week 28 vs week 52). Assess if epigenetic age could be a marker for the effect of tildrakizumab on psoriasis through psoriasis severity scores.

Specific Aim 3: We will evaluate the transcriptomic impact of ILUMYA therapy in patients with psoriasis and possible correlation/association with Epigenetic changes, psoriasis severity scores, the presence of systemic comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Age: 35 years of age or older.
* Psoriasis subjects: moderate-to-severe psoriasis: PASI (Psoriasis Area and Severity Index ≥12) and a minimum Body Surface Area (BSA) involvement of 10%.
* Control Subjects: other skin diseases without psoriasis.

Exclusion Criteria:

1. Patients aged less than 35 years.
2. Patients with previous skin cancer or other cancers.
3. Women of childbearing potential without effective contraceptive method, or lactating women.
4. Prisoners.
5. Psoriasis patients who have had a severe allergic reaction to ILUMYA or any of its ingredients.
6. Psoriasis patients who have chronic or recurring infections. Positive QuantiFERON upon screening will be exclusionary for this trial (latent tuberculosis).
7. Any condition that, in the opinion of the investigator, may interfere with patient's ability to participate in the study, such as severe cognitive impairment or other comorbidities that would, in the opinion of the investigator, predictably limit compliance with the study plan.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Epigenetic aging in psoriatic patients. | Baseline
  To examine the association between epigenetic age acceleration and psoriasis: by comparing the baseline samples of peripheral blood leukocyte genome-wide DNA methylation assay sample collected at the screening visit for psoriasis vs non-psoriasis patients.
  The epigenetic aging test is based on the Methylation EPIC BeadChip (Illumina), covering over 850,000 methylation sites. Specific patterns and quantifications will be compared between groups.
Dynamics of tildrakizumab on epigenetic aging of psoriatic patients. | Baseline and treatment weeks 28 and 52.
  To evaluate dynamic effects and changes in epigenetic age of the on-label use of ILUMYA (week 28 vs screening visit). And upon discontinuation (week 28 vs week 52). Assess if epigenetic age could be a marker for the effect of ILUMYA on psoriasis through psoriasis severity scores.
  Specific patterns and quantifications will be compared between timeframes.

SECONDARY OUTCOMES:
Evaluate the transcriptomic impact of tildrakizumab therapy in patients with psoriasis | Baseline and treatment week 28.
  To evaluate the blood transcriptome changes with anti-IL-23 therapy in patients with psoriasis, and possible correlation/association with psoriasis severity scores (BSA, PASI and CAPP), serum markers, and the presence of systemic co-morbidities on epigenetic aging.
Effects of individual characteristics on tildrakizumab response | Baseline and treatment weeks 28 and 52.
  To evaluate the possible correlation/association with changes in psoriasis severity scores (BSA, PASI and CAPP) and the presence of systemic co-morbidities on epigenetic aging. Multivariate analysis will be conducted with variables that include, but are not limited to baseline epigenetic aging assay results, age, body mass index, previous diagnoses, and medical interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos G Wambier, MD, PhD, Principal Investigator — Department of Dermatology, Warren Alpert Medical School of Brown University
Locations (1):
- Clinical Trials Center for Skin Diseases: Rhode Island Hospital, 593 Eddy Street, Dermatology Research, Jane Brown Building, 1st floor, Room 115, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lowes MA, Bowcock AM, Krueger JG. Pathogenesis and therapy of psoriasis. Nature. 2007 Feb 22;445(7130):866-73. doi: 10.1038/nature05663. PMID 17314973
- [Background] Kurd SK, Gelfand JM. The prevalence of previously diagnosed and undiagnosed psoriasis in US adults: results from NHANES 2003-2004. J Am Acad Dermatol. 2009 Feb;60(2):218-24. doi: 10.1016/j.jaad.2008.09.022. Epub 2008 Nov 20. PMID 19022533
- [Background] Li WQ, Cho E, Weinstock MA, Mashfiq H, Qureshi AA. Epidemiological Assessments of Skin Outcomes in the Nurses' Health Studies. Am J Public Health. 2016 Sep;106(9):1677-83. doi: 10.2105/AJPH.2016.303315. Epub 2016 Jul 26. PMID 27459457
- [Background] Li W, Han J, Hu FB, Curhan GC, Qureshi AA. Psoriasis and risk of type 2 diabetes among women and men in the United States: a population-based cohort study. J Invest Dermatol. 2012 Feb;132(2):291-8. doi: 10.1038/jid.2011.319. Epub 2011 Oct 13. PMID 21993559
- [Background] Li WQ, Han JL, Manson JE, Rimm EB, Rexrode KM, Curhan GC, Qureshi AA. Psoriasis and risk of nonfatal cardiovascular disease in U.S. women: a cohort study. Br J Dermatol. 2012 Apr;166(4):811-8. doi: 10.1111/j.1365-2133.2011.10774.x. PMID 22175820
- [Background] Li WQ, Han JL, Chan AT, Qureshi AA. Psoriasis, psoriatic arthritis and increased risk of incident Crohn's disease in US women. Ann Rheum Dis. 2013 Jul;72(7):1200-5. doi: 10.1136/annrheumdis-2012-202143. Epub 2012 Aug 31. PMID 22941766
- [Background] Merola JF, Wu S, Han J, Choi HK, Qureshi AA. Psoriasis, psoriatic arthritis and risk of gout in US men and women. Ann Rheum Dis. 2015 Aug;74(8):1495-500. doi: 10.1136/annrheumdis-2014-205212. Epub 2014 Mar 20. PMID 24651620
- [Background] Ryan C, Korman NJ, Gelfand JM, Lim HW, Elmets CA, Feldman SR, Gottlieb AB, Koo JY, Lebwohl M, Leonardi CL, Van Voorhees AS, Bhushan R, Menter A. Research gaps in psoriasis: opportunities for future studies. J Am Acad Dermatol. 2014 Jan;70(1):146-67. doi: 10.1016/j.jaad.2013.08.042. Epub 2013 Oct 11. PMID 24126079
- [Background] Gudjonsson JE, Krueger G. A role for epigenetics in psoriasis: methylated Cytosine-Guanine sites differentiate lesional from nonlesional skin and from normal skin. J Invest Dermatol. 2012 Mar;132(3 Pt 1):506-8. doi: 10.1038/jid.2011.364. PMID 22327261
- [Background] Nelson HH, Kelsey KT. Epigenetic epidemiology as a tool to understand the role of immunity in chronic disease. Epigenomics. 2016 Aug;8(8):1007-9. doi: 10.2217/epi-2016-0055. Epub 2016 Jul 13. No abstract available. PMID 27411030
- [Background] Horvath S. DNA methylation age of human tissues and cell types. Genome Biol. 2013;14(10):R115. doi: 10.1186/gb-2013-14-10-r115. PMID 24138928
- [Background] Bocklandt S, Lin W, Sehl ME, Sanchez FJ, Sinsheimer JS, Horvath S, Vilain E. Epigenetic predictor of age. PLoS One. 2011;6(6):e14821. doi: 10.1371/journal.pone.0014821. Epub 2011 Jun 22. PMID 21731603
- [Background] Hannum G, Guinney J, Zhao L, Zhang L, Hughes G, Sadda S, Klotzle B, Bibikova M, Fan JB, Gao Y, Deconde R, Chen M, Rajapakse I, Friend S, Ideker T, Zhang K. Genome-wide methylation profiles reveal quantitative views of human aging rates. Mol Cell. 2013 Jan 24;49(2):359-367. doi: 10.1016/j.molcel.2012.10.016. Epub 2012 Nov 21. PMID 23177740
- [Background] Marioni RE, Shah S, McRae AF, Chen BH, Colicino E, Harris SE, Gibson J, Henders AK, Redmond P, Cox SR, Pattie A, Corley J, Murphy L, Martin NG, Montgomery GW, Feinberg AP, Fallin MD, Multhaup ML, Jaffe AE, Joehanes R, Schwartz J, Just AC, Lunetta KL, Murabito JM, Starr JM, Horvath S, Baccarelli AA, Levy D, Visscher PM, Wray NR, Deary IJ. DNA methylation age of blood predicts all-cause mortality in later life. Genome Biol. 2015 Jan 30;16(1):25. doi: 10.1186/s13059-015-0584-6. PMID 25633388
- [Background] Christiansen L, Lenart A, Tan Q, Vaupel JW, Aviv A, McGue M, Christensen K. DNA methylation age is associated with mortality in a longitudinal Danish twin study. Aging Cell. 2016 Feb;15(1):149-54. doi: 10.1111/acel.12421. Epub 2015 Nov 17. PMID 26594032
- [Background] Horvath S, Erhart W, Brosch M, Ammerpohl O, von Schonfels W, Ahrens M, Heits N, Bell JT, Tsai PC, Spector TD, Deloukas P, Siebert R, Sipos B, Becker T, Rocken C, Schafmayer C, Hampe J. Obesity accelerates epigenetic aging of human liver. Proc Natl Acad Sci U S A. 2014 Oct 28;111(43):15538-43. doi: 10.1073/pnas.1412759111. Epub 2014 Oct 13. PMID 25313081
- [Background] Horvath S, Ritz BR. Increased epigenetic age and granulocyte counts in the blood of Parkinson's disease patients. Aging (Albany NY). 2015 Dec;7(12):1130-42. doi: 10.18632/aging.100859. PMID 26655927
- [Background] Horvath S, Levine AJ. HIV-1 Infection Accelerates Age According to the Epigenetic Clock. J Infect Dis. 2015 Nov 15;212(10):1563-73. doi: 10.1093/infdis/jiv277. Epub 2015 May 12. PMID 25969563
- [Background] Levine ME, Hosgood HD, Chen B, Absher D, Assimes T, Horvath S. DNA methylation age of blood predicts future onset of lung cancer in the women's health initiative. Aging (Albany NY). 2015 Sep;7(9):690-700. doi: 10.18632/aging.100809. PMID 26411804
- See also: Brown Dermatology Clinical Trials Website — https://brownderm.org/clinical-trials/